CLINICAL TRIAL: NCT04626804
Title: Remember Stuff: A Dyadic-focused Technology to Support Persons With Alzheimer's Disease in the Community
Acronym: R/S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Nicole R. Fowler, PhD, Associate Professor of Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2006294326
Record Dates: First submitted 2020-11-03; First posted 2020-11-13 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Anxiety; Depression; Caregiver Burnout; Anxiety Generalized
Keywords: Alzheimer's disease; Dementia; Caregiving; Caregiver; Anxiety; Telehealth
MeSH Terms: conditions — Anxiety Disorders; Depression; Caregiver Burden; Generalized Anxiety Disorder; Alzheimer Disease; Dementia | interventions — Amyloid beta-Protein Precursor

STUDY DESIGN:
Intervention Model Description: single dyadic group focused on determining acceptance and feasibility of the in home computer monitor individually programmed for each dyadic needs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 Test the usability, perceptions, and acceptability of R/S (Experimental): Dyads will use the R/S unit for 90 days, unless they request it to be removed prior to the end of the study. . The primary outcome is a caregiver-assessed measure usability.
  Interventions: Other: Remember Stuff: A Dyadic-focused Technology to Support Persons with Alzheimer's Disease in the Community

INTERVENTIONS:
Other: Remember Stuff: A Dyadic-focused Technology to Support Persons with Alzheimer's Disease in the Community — testing the usability, perceptions, and acceptability of R/S among dyads of older adults with early Alzheimer's disease and other related dementias
  Other Names: System Usability Scale; Participant Willingness to Use; The Behavioral Intention Scale; Performance Expectancy; Computer Literacy

SUMMARY:
Test the usability, perceptions and acceptability of a computer monitor for participant diagnosed with ADRD and their caregiver who will program the applications specifically for each individual to help them remember activities of daily living. Goal is to keep participants in their homes longer and delay the need for institutional care

DETAILED DESCRIPTION:
Dyads will use the R/S unit for 90 days, unless they request it to be removed prior to the end of the study. The research team (N. Fowler, PhD) will assess measures at baseline, 30 days, 60 days and 90 days. The primary outcome is a caregiver-assessed measure usability. Secondary measures include patient- assessed usability, and objective measures of frequency and type of use and computer literacy for both caregiver and the individual with ADRD22. Methods to collect user data (frequency, clicks, etc.) will be collected using tools developed in Aim 2. Desired outcome measures include (1) a mean score of >80 ("Good") on the ten-item System Usability Scale (SUS) modified by IU investigators to accommodate older adults23; (2) a 80 percent acceptability rate on the Behavioral Intention 3-item scale; and, (3) at least 70 percent of participants using R/S a minimum of weekly. SUS is a validated ten-item scale (e.g., "Learning to use RememberStuff® was quick for me") using a five-point response scale (strongly disagree to strongly agree). Acceptance will be assessed as the mean score on a 3-item Satisfaction scale (e.g., "Rate your satisfied with RememberStuff®?"). This scale was adapted by IU Investigators for health IT and uses a seven-point response scale from 0 (not at all) to 6 (a great deal). Satisfaction is one of the canonical assessments for user acceptance of technology. SUS and Satisfaction questionnaires will be researcher-administered by study staff either face-to-face in the participant's homes, or via telephone. The mean and standard deviation for the composite SUS, acceptability rate and weekly usage will be calculated to a 90% confidence interval. Other secondary measures are adapted from Holden et al and are guided by the UTAUT221. Mean caregiver scores on the measures will also be compared to mean scores of the patient measures to examine congruence in usability and acceptability within the dyad.

ELIGIBILITY:
Patient Inclusion Criteria:

* achieve a Montreal Cognitive Assessment (MoCA) score of 6-17 (mild to moderate dementia)
* diagnosis of early Alzheimer's disease or related dementia or caregiver reports ADRD diagnosis (if community based recruitment)
* provide identification of a caregiver (living with or otherwise involved in the ongoing care of the person with ADRD)
* able to communicate in English
* able to provide informed consent

Patient Exclusion Criteria:

* lives in a nursing home or long term care facility or assisted living facility
* do not pass the MoCA with a score between 6-17
* unable to identify a caregiver
* is limited by severe arthritis or other condition in the use of his/her hands

Caregiver Inclusion Criteria:

* 21 years or older
* able to provide informed consent
* able to communicate in English

Caregiver Exclusion Criteria:

* under 21 years of age
* does not have access to a computer/device
* diagnosis of ADRD
* diagnosis of serious mental illness (i.e. schizophrenia)

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Usability | through study completion, an average of 4 months
  Satisfaction and use of the monitor and apps using the Usability Scale, a validated 10-item scale sithe items suchs as "learning to use the calendar function was quick for me", using a 5 point response scale (0= strongly disagree to 5= strongly agree)
  Usability Scale, a validated 10-item scale (e.g. "Learning to use Calendar function was quick for me" using a 5-point response scale (0=strongly disagree to 5= strongly agree)

SECONDARY OUTCOMES:
Acceptability | through study completion, an average of 4 months
  Acceptability satisfaction assessed by the VAS using a 3-item score: participants willingness to use "Assuming I have access to this technology today, I would use it". Participants' willingness to use in the future "I could imagine using this technology in the future". Perceived usefulness scale -Using this technology would be a relief for my daily care routine. "Altogether I think this technology would be useful in my daily care routine. Perecived ease of use scale- Interacting with the technology would not require a lot of mental effort "I think I would have the technology under control- Altogether I think the technology would be easy to use".
Intention of Use | through study completion, an average of 4 months
  The Behavioral Intention scale (e.g., "If it were up to you, to what extent would you want to use RememberStuff®?"). The 4-item scale uses a 7-point response scale from 0 (not at all) to 6 (a great deal). Behavioral intention is the canonical assessment for user acceptance of technology
Performance expectancy | through study completion, an average of 4 months
  7 items (e.g. "Thinking about using RememberStuff® in the past 90 days, to what extent do you find it useful in your daily life?") that use a 7-point response scale from 0 (not at all) to 6 (a great deal). 3-5 Semi-structured and open-ended questions about experience using the technology.
Computer literacy | through study completion, an average of 4 months
  The Computer Literacy Scale for Older Adults-12 (CLS-12)24 is a validated measure that assess frequency of 11 different computer related tasks including knowledge of symbols, terms related to computers and electronic devices, and internet use

OTHER OUTCOMES:
Dementia Severity Scale | through study completion, an average of 4 month
  validated tool measuring dementia severity at specific intervals of the study

CONTACTS AND LOCATIONS:
Overall Officials: Nicole R Fowler, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
In future manuscripts, the authors will list contact information and state that the IPD is available upon request
Time Frame: at the completion of the study, within 12 months
Access Criteria: at the completion of the study, within 12 months